CLINICAL TRIAL: NCT06744504
Title: Anthracycline-based Standard-dose vs Intermediate-dose Cytarabine Induction in the Treatment of Acute Myeloid Leukemia With RUNX1-RUNX1T1: a Prospective, Randomized, Controlled Phase III Clinical Trial
Brief Title: Standard-dose vs Intermediate-dose Cytarabine Induction in the Treatment of Acute Myeloid Leukemia With RUNX1-RUNX1T1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024094
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-11

CONDITIONS: AML; RUNX1-RUNX1T1 Fusion Protein Expression
MeSH Terms: interventions — Cytarabine; Daunorubicin; Idarubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard-dose Cytarabine (Active Comparator): Induction therapy:
  Cytarabine (Ara-c) 100mg/ m2/ day, day 1-7; Daunorubicin (DNR) 60mg/m2/ day, day 1-3; Those who did not meet CR were treated with IAC regimen.
  IAC:
  IDA 8 mg/m2/d, D1-3; Ara-c 100 mg/m2, D1-7; CTX 350mg/m2, D2,5;
  Post-remission treatment options:
  High dose Ara-C(HDAC) : 3 cycles Ara-C 3g/㎡/q12h, days 1, 3 and 5 For patietns RUNX1-RUNX1 MRD reduction < 3 logs after 2 courses, allo-transplantation is recommended if donor is available.
  Interventions: Drug: cytarabine; Drug: daunorubicin; Drug: idarubicin; Drug: cyclophosphamide
- Intermediate-dose Cytarabine (Experimental): Induction therapy:
  Cytarabine (Ara-c) 100mg/ m2/ day, day 1-4; 1g/㎡/q12h, day 5-7; Daunorubicin (DNR) 60mg/m2/ day, day 1-3; Those who did not meet CR were treated with IAC regimen.
  IAC:
  IDA 8 mg/m2/d, D1-3; Ara-c 100 mg/m2, D1-7; CTX 350mg/m2, D2,5;
  Post-remission treatment options:
  High dose Ara-C(HDAC) : 3 cycles; Ara-C 3g/㎡/q12h, days 1, 3 and 5. For patietns RUNX1-RUNX1 MRD reduction < 3 logs after 2 courses, allo-transplantation is recommended if donor is available.
  Interventions: Drug: cytarabine; Drug: daunorubicin; Drug: idarubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: cytarabine — Cytarabine combined with daunorubicin was used for induction therapy. According to the different doses of cytarabine, it was divided into standard dose group and intermediate dose group.In addition, high doses of cytarabine are also used for post-remission treatment.
Drug: daunorubicin — combined with cytarabine and used for induction therapy
Drug: idarubicin — combined with cytarabine and cyclophosphamide and used for post-remission treatment
Drug: cyclophosphamide — combined with cytarabine and idarubicin and used for post-remission treatment

SUMMARY:
Leukemia is one of the common malignant tumors that threaten human health. Although the efficacy of AML treatment has improved significantly in recent years, it remains one of the major diseases threatening human health. Current research on AML treatment mainly has two directions. One is the addition of new targeted therapy drugs, and the other research direction is to enhance the intensity of AML chemotherapy, including the use of large doses of anthracycline drugs or the use of high-dose cytarabine treatment.

Since the 1990s, induction remission has been achieved by using anthracyclines in combination with high-dose cytarabine. The ECOG (Eastern Cooperative Oncology Group) contends that high-dose induction chemotherapy fails to enhance the bone marrow remission rate but elevates the chemotherapy-related mortality rate. Bradstock and the Australian Group also noted that although it does not increase the bone marrow remission rate, it can result in longer survival time and disease-free survival time. The clinical study from EORTC-GIMEMA AML-12 discovered that AML patients under the age of 45 could benefit from induction therapy incorporating high-dose cytarabine. In our previous randomized controlled clinical trials, it was found that the HAD and DA regimens containing intermediate-dose cytarabine could enhance the complete remission rate and improve the overall survival of adult AML. However, the degree of benefit varies among different AML subgroups.

The abnormalities of RUNX1-RUNX1T1 and CBFβ-MYH11 respectively involve a subunit of CBF (core binding factor), thus the two are collectively called CBF leukemia. Previous retrospective studies show that this type of leukemia benefits from intensified treatment regimens such as FLAG. However, at present, there is a lack of prospective randomized controlled clinical studies to confirm this. Therefore, in this study, we intend to further verify through a prospective randomized controlled clinical trial whether the induction treatment regimen containing intermediate-dose cytarabine can improve the long-term efficacy of adult RUNX1-RUNX1T1 acute myeloid leukemia.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled phase III clinical trial that plans to enroll adult patients with AML who meet the WHO (2022) or ICC criteria for eligibility for intensive chemotherapy with RUNX1-RUNX1 fusion. For patients who meet the inclusion criteria and do not meet any exclusion criteria, they will be randomly assigned to either the A group, which receives standard-dose DA induction therapy, or the B group, which receives intermediate-dose DA induction therapy. Patients who do not achieve complete remission after one cycle of induction therapy will receive IAC reinduction therapy. Patients who achieve complete remission after one or two cycles of induction therapy will proceed to receive three cycles of high-dose cytarabine consolidation therapy. Patients who do not achieve complete remission after two cycles of induction therapy will be withdrawn from the treatment protocol. For patients whose fusion gene levels do not meet the criteria, allogeneic hematopoietic stem cell transplantation is recommended.

ELIGIBILITY:
Inclusion Criteria:

1. AML conforming to WHO (2022) or ICC standards
2. Possessing the RUNX1::RUNX1T1 fusion gene
3. Age ranging from 14 to 60 years old, regardless of gender.
4. The performance status assessment of the Eastern Cooperative Oncology Group (ECOG-PS) being 0 - 2.
5. Meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment):

1) Total bilirubin ≤ 1.5 times the upper limit of the normal value for the same age group; 2) AST and ALT ≤ 2.5 times the upper limit of the normal value for the same age group; 3) Serum creatinine < 2 times the upper limit of the normal value for the same age group; 4) Cardiac enzymes < 2 times the upper limit of the normal value for the same age group; 5) The cardiac ejection fraction determined by echocardiography (ECHO) > 50%. An informed consent form must be signed before the commencement of all specific research procedures, either by the patient themselves or their immediate relatives. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the disease, the informed consent form shall be signed by the legal guardian or the immediate relatives of the patient.

Exclusion Criteria:

1. Acute promyelocytic leukemia accompanied by PML-RARA fusion gene.
2. Acute myeloid leukemia featuring BCR-ABL fusion gene.
3. Patients undergoing retreatment (but can receive cytoreductive therapy with hydroxyurea and cytarabine).
4. Individuals concurrently having malignant tumors in other organs (requiring treatment).
5. Active cardiac disorders, defined as one or more of the following:

1) A history of uncontrolled or symptomatic angina pectoris; 2) Myocardial infarction less than 6 months from study enrollment; 3) A history of significant arrhythmia requiring medication or presenting with severe clinical symptoms; 4) Uncontrolled or symptomatic congestive heart failure (> NYHA Class 2)

6. Severe infectious diseases (untreated tuberculosis, pulmonary aspergillosis).

7. Individuals deemed ineligible for enrollment by the investigator.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 2 years after the date of the last enrolled participants
  Used to evaluate all patients who enter clinical trials. From the date of entry into the trial until the date of patient death (including any cause) or last survival follow-up.

SECONDARY OUTCOMES:
Complete remission (CR)/CR with partial hematologic recovery (CRh)/CR with incomplete hematologic recovery (CRi) rate after induction therapy | up to 3 months after the date of the last enrolled participants
  The ratio of patients achieved CR/CRh/CRi after induction therapy.
RUNX1::RUNX1T1 minimal residual disease (MRD) reduction >3 logs after 2 courses | up to 2 years after the date of the last enrolled participants
  RUNX1::RUNX1T1 MRD is measured by real-time PCR.
RUNX1::RUNX1T1 molecular MRD undectable rate | up to 2 years after the date of the last enrolled participants
  MRD levels monitored by polymerase chain reaction are associated with outcomes in acute myeloid leukemia with RUNX1-RUNX1T1.
Relapse-free survival (RFS) | up to 2 years after the date of the last enrolled participants
  Defined only for patients achieving CRc; measured from the date of achievement of remission until the date of hematologic relapse or death from any cause; patients not known to have relapsed or died at last follow-up are censored on the date they were last known to be alive
Event-free survival (EFS) | up to 2 years after the date of the last enrolled participants
  All patients definitions for the trial; From the date of enrollment to the time of treatment failure after two courses of induction therapy, recurrence after CRc, date of all-cause death, or the date of last survival follow-up.
30-day mortality | within 30 days of the date of the last enrolled participants
  Percentage of patients who died within 30 days from enrollment.
60-day mortality | within 60 days of the date of the last enrolled participants
  Percentage of patients who died within 60 days from enrollment
Complete remission (CR)/CR with partial hematologic recovery (CRh)/CR with incomplete hematologic recovery (CRi) rate | up to12 months after the date of the last enrolled participants
  the ratio of patients achieved CR/CRh/CRi

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No